CLINICAL TRIAL: NCT00757523
Title: A Multi-center, Randomized, Evaluator-blind, Parallel-group Evaluation of the Efficacy, Safety, and Tolerability of Duac Akne Gel and Epiduo Gel in the Topical Treatment of Facial Acne Vulgaris
Brief Title: Evaluation of the Effectiveness, Safety, and Tolerability of Duac Akne Gel and Epiduo Gel in the Treatment of Facial Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S194-401
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Akne; Acne; Akne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epiduo Gel (Active Comparator): Epiduo Gel (combination of 0.1% adapalene and 2.5% benzoyl peroxide (BPO) in a gel preparation).
  Interventions: Drug: Epiduo Gel
- Duac Gel (Experimental): Duac Akne Gel (combination of 1% clindamycin phosphate and 5% benzoyl peroxide (BPO) in a gel preparation).
  Interventions: Drug: Duac Gel

INTERVENTIONS:
Drug: Epiduo Gel — Epiduo Gel (combination of 0.1% adapalene and 2.5% benzoyl peroxide (BPO) in a gel preparation). Treatments administered once-daily in the evening for 12 weeks
  Arms: Epiduo Gel
Drug: Duac Gel — Duac Akne Gel (combination of 1% clindamycin phosphate and 5% benzoyl peroxide (BPO) in a gel preparation). Treatments administered once-daily in the evening for 12 weeks
  Other Names: Duac Akne Gel
  Arms: Duac Gel

SUMMARY:
The purpose of this study is to compare the effectiveness of two marketed products in subjects with facial acne vulgaris

DETAILED DESCRIPTION:
Multiple physiopathological factors have been associated with acne vulgaris. Drug combinations are frequently used to address these factors and to improve efficacy in the treatment of acne. The current study proposes to compare a fixed-dose (once-daily) combination gel product containing benzoyl peroxide (BPO)and clindamycin against a fixed-dose (once-daily) combination gel product containing BPO and adapalene for the treatment of facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12 to 45 years of age, inclusive, in good general health.
* Clinical diagnosis of acne vulgaris
* Capable of understanding and willing to provide signed and dated written voluntary informed consent
* Female subjects of childbearing potential must have a negative pregnancy test at baseline. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception
* Subjects who have been treated with estrogens, androgens, or anti-androgenic agents for more than 12 consecutive weeks prior to the first dose of study product are allowed to enroll as long as they do not expect to change dose, drug, or discontinue use during the study.
* The ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.

Exclusion Criteria:

* Female subjects who are pregnant, trying to become pregnant, or who are lactating.
* Any clinically relevant finding at their baseline physical examination or medical history such as severe systemic diseases or diseases of the facial skin other than acne vulgaris.
* Facial hair that may obscure the accurate assessment of acne grade.
* History or presence of regional enteritis or inflammatory bowel disease (eg, ulcerative colitis, pseudomembranous colitis, chronic diarrhea, or a history of antibiotic-associated colitis) or similar symptoms.
* Used topical antibiotics on the face or systemic antibiotics within the past 2 and 4 weeks, respectively.
* Used topical corticosteroids on the face or systemic corticosteroids within the past 4 weeks. Use of inhaled, intra articular or intra-lesional (other than for facial acne lesions) steroids is acceptable.
* Used systemic retinoids within the past 6 months.
* Using drugs known to be photosensitizers (eg, thiazides, tetracyclines, fluoroquinolones, phenothiazines, sulfonamides) because of the possibility of increased phototoxicity.
* Using neuromuscular blocking agents. Clindamycin has neuromuscular blocking activities, which may enhance the action of other neuromuscular blocking agents.
* Used topical anti-acne medications (eg, BPO, retinoids, azelaic acid, resorcinol, salicylates, sulfacetamide sodium and derivatives, glycolic acid) within the past 2 weeks.
* Used any investigational therapy within 4 weeks of study day 1.
* Using the following types of facial products: astringents, toners, abradants, facials, peels containing glycolic or other acids, masks, washes or soaps containing BPO, sulfacetamide sodium or salicylic acid, non-mild facial cleansers, or moisturizers that contain retinol, salicylic acid, or α- or β-hydroxy acids.
* Using medications that are reported to exacerbate acne (eg, mega-doses of certain vitamins such as vitamin D, vitamin A, and vitamins B2, B6, and B12; haloperidol; halogens such as iodide and bromide; lithium; hydantoin; and phenobarbital) as these may impact efficacy assessments.
* Have had a facial procedure (chemical or laser peel, microdermabrasion, artificial ultraviolet [UV] therapy) performed by an esthetician, beautician, physician, nurse, or other practitioner, within the past 4 weeks.
* Have a known hypersensitivity or previous allergic reaction to any of the active components, lincomycin, adapalene, clindamycin, BPO, or excipients of the study medication.
* Employees of a clinical research organization involved in the study, or Stiefel Laboratories, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee.
* Have a member of the same household in this trial.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2008-09-10 (Actual); Primary Completion 2009-04-24 (Actual); Study Completion 2009-06-24 (Actual)

PRIMARY OUTCOMES:
Percent change in inflammatory lesion count from Baseline to Week 12 | Baseline (Day 1) and Week 12
  The efficacy assessor performed a count of inflammatory lesions (papules and pustules, including nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Week 12.

SECONDARY OUTCOMES:
Percentage of participants who achieved treatment success, defined as improvement of 2 grades or more in their Investigator Static Global Assessment (ISGA) acne severity scale from Baseline to Week 12 | Week 12
  ISGA success was defined as the improvement of 2 grades or more in the participant's acne severity scale at Week 12. The area considered for assessment must be confined to the face. Acne severity of the participant's face was assessed by the assessor using the ISGA scale, ranging from 0 to 5 where 0=Clear skin with no inflammatory or non-inflammatory lesions. ;1=almost clear: Rare non-inflammatory lesions with no more than one small inflammatory lesion ;2=mild: Some non-inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions). ;3=moderate: Up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion; 4=severe: Up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions and 5= Very Severe: Many non-inflammatory and inflammatory lesions and more than a few nodular lesions. May have cystic lesions. The higher score indicated more severe lesions.
Time to 2-grade improvement in ISGA from Baseline | Week 12
  ISGA success was defined as the improvement of 2 grades or more in the participant's acne severity scale at Week 12. Time to ISGA success from Baseline was analyzed using Kaplan-Meier Estimate of time. Baseline was defined as the value at Day 1 (Visit 1). Participants with missing week 12 evaluations were considered failures.
Percent change in total lesion count from Baseline to week 12 | Baseline (Day 1) and Week 12
  The efficacy assessor performed a count of total lesions at each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Week 12.
Absolute change in inflammatory lesion count from Baseline to Weeks 1, 2, 4, 8 | Baseline (Day 1) and Weeks 1, 2, 4, 8
  The efficacy assessor performed a count of inflammatory lesions (papules and pustules, including nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Weeks 1, 2, 4, 8.
Absolute change in inflammatory lesion count from Baseline to Week 12. | Baseline (Day 1) and Week 12
  The efficacy assessor performed a count of inflammatory lesions (papules and pustules, including nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Week 12.
Absolute change in total lesion count from Baseline to Weeks 1, 2, 4, 8 | Baseline (Day 1) and Weeks 1, 2, 4, 8
  The efficacy assessor performed a count of total lesions at each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Weeks 1, 2, 4, 8.
Absolute change in total lesion count from Baseline to Week 12 | Baseline (Day 1) and Week 12
  The efficacy assessor performed a count of total lesions at each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Week 12.
Percentage of participants who achieved treatment success from Baseline to Weeks 1, 2, 4, and 8 | Weeks 1, 2, 4, and 8
  ISGA success was defined as the improvement of 2 grades or more in the participant's acne severity scale at Week 12. Acne severity of the participant's face was assessed by the assessor using the ISGA scale, ranging from 0 to 5 where 0= Clear skin with no inflammatory or non-inflammatory lesions and 5= Very Severe: Many non-inflammatory and inflammatory lesions and more than a few nodular lesions. May have cystic lesions. The higher score indicated more severe lesions. The area considered for the ISGA was confined to the face. Data for percentage of participants who achieved treatment success from Baseline to Weeks 1, 2, 4, and 8 was not collected.
Absolute change in non-inflammatory lesion count from Baseline to Weeks 1 2, 4,8 | Baseline (Day 1) and Weeks 1,2,4,8
  The efficacy assessor performed a count of non-inflammatory lesions (open and closed comedones, excluding nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Weeks 1, 2, 4, 8.
Absolute change in non-inflammatory lesion count from Baseline to Week 12 | Baseline (Day 1) and Week 12
  The efficacy assessor performed a count of non-inflammatory lesions (open and closed comedones, excluding nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Week 12.
Percent change in non-inflammatory lesion count from Baseline to Weeks 1, 2, 4, 8 | Baseline (Day 1) and Weeks 1, 2, 4, 8
  The efficacy assessor performed a count of non-inflammatory lesions (open and closed comedones, excluding nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Weeks 1, 2, 4, 8.
Percent change in non-inflammatory lesion count from Baseline to Week 12 | Baseline (Day 1) and Week 12
  The efficacy assessor performed a count of non-inflammatory lesions (open and closed comedones, excluding nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Week 12.
Percent change in inflammatory lesion count from Baseline to Weeks 1, 2, 4, and 8 | Baseline (Day 1) and Weeks 1, 2, 4, and 8
  The efficacy assessor performed a count of inflammatory lesions (papules and pustules, including nasal lesions) each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Weeks 1, 2, 4, and 8.
Percent change in total lesion count from Baseline to Weeks 1, 2, 4, and 8 | Baseline (Day 1) and Weeks 1, 2, 4, and 8
  The efficacy assessor performed a count of total lesions at each study visit. Lesion counts were confined to the face. Baseline was defined as the value at Day 1 (Visit 1). Change from Baseline was calculated by subtracting the Baseline from the post-randomization value at Weeks 1, 2, 4, and 8.
Time to reach 50 percent reduction in inflammatory lesion counts from Baseline | Week 12
  Time to reach 50 percent reduction in inflammatory lesion counts (papules and pustules, including nasal lesions) from Baseline was analyzed using Kaplan-Meier Estimate of time. Baseline was defined as the value at Day 1 (Visit 1).
Time to reach 50 percent reduction in non-inflammatory lesion counts from Baseline | Week 12
  Time to reach 50 percent reduction in non-inflammatory lesion counts ((open and closed comedones, excluding nasal lesions) from Baseline was analyzed using Kaplan-Meier Estimate of time. Baseline was defined as the value at Day 1 (Visit 1).
Time to reach 50 percent reduction in total lesion counts from Baseline | Week 12
  Time to time to reach 50 percent reduction in total lesion counts from Baseline was analyzed using Kaplan-Meier Estimate of time. Baseline was defined as the value at Day 1 (Visit 1).
Percentage of participants who had a Subject's Global Change Assessment score (SGAC) of 0 or 1 at Weeks 1, 2, 4, 8, and 12 | Upto Week 12
  SGCA is measured on a scale (Clear, Almost Clear, Mild, Moderate, Severe, Very Severe) with Clear being best and Very Severe being worst. The area considered for the ISGA was confined to the face. Data for percentage of participants who had a SGAC of 0 or 1 at Weeks 1, 2, 4, 8, and 12 was not collected.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Germany (15):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Dessau
  - GSK Investigational Site, Dülmen
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Giessen
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Kiel
  - GSK Investigational Site, Landau
  - GSK Investigational Site, Magdeburg
  - GSK Investigational Site, München
  - GSK Investigational Site, Münster
  - GSK Investigational Site, Potsdam

REFERENCES:
- [Result] Zouboulis CC, Fischer TC, Wohlrab J, Barnard J, Alio AB. Study of the efficacy, tolerability, and safety of 2 fixed-dose combination gels in the management of acne vulgaris. Cutis. 2009 Oct;84(4):223-9. PMID 19911678